CLINICAL TRIAL: NCT03990480
Title: Valsartan Versus Amlodipine Effect on Left Ventricular Multidirectional Deformation and Adipocytokines Level in Hypertensive Patients: Speckle Tracking Echocardiography
Brief Title: Valsartan Versus Amlodipine Effect on Left Ventricular Multidirectional Deformation and Adipocytokines Level
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Clinical Pharmacy Lecturer, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Valsartan versus Amlodipine LV
Record Dates: First submitted 2019-06-16; First posted 2019-06-19 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Amlodipine

STUDY DESIGN:
Intervention Model Description: Thirty control healthy individuals and 200 patients with uncomplicated, essential hypertension were enrolled and followed up for 3 months in a controlled randomized study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- valsartan (Active Comparator): Group I treated with valsartan (160 mg/d, n = 100)
  Interventions: Drug: valsartan (160 mg/d)
- amlodipine (Active Comparator): Group II amlodipine (10 mg/d, n = 100).
  Interventions: Drug: amlodipine (10 mg/d).
- Control (No Intervention): 30 healthy subjects are enrolled as control group (Group III).

INTERVENTIONS:
Drug: valsartan (160 mg/d) — Group I treated with valsartan (160 mg/d, n = 100)
  Other Names: Tareg 160 mg
  Arms: valsartan
Drug: amlodipine (10 mg/d). — Group II amlodipine (10 mg/d, n = 100).
  Other Names: Norvasc 10 mg
  Arms: amlodipine

SUMMARY:
Aim: To evaluate the effects of Valsartan versus Amlodipine on LV deformation in relation to plasma adiponectin and leptin levels in hypertensive individuals.

Methods: LV strain measured by 2 dimensional speckle tracking echocardiography, plasma levels of adiponectin and leptin was determined in 30 healthy individuals served as control group and in 200 hypertensive patients before and after treatment for three months with either Valsartan 160 mg or amlodipine 10 mg.

DETAILED DESCRIPTION:
Patients and methods Thirty control healthy individuals and 200 patients with uncomplicated, essential hypertension were enrolled and followed up for 3 months in a controlled randomized study. All subjects' health status was evaluated by a complete medical examination. All BP measurements were made with calibrated mercury manometers (Korotkoff I and V). Three separate measurements were taken at least 2 min apart and the average of these values was calculated. Subjects' height and weight were recorded in the fasting state with the subjects wearing only light clothes and without shoes and BMI was calculated using the equation (BMI = weight (kg)/height (m)2). Patients, of both sexes with mild to moderate essential hypertension (diastolic blood pressure [DBP] >80 and ≤100 mmHg after a 2-week wash-out period, SBP systolic blood pressure>120 and 160 mmHg). Patients were randomly assigned into two groups using a computer-generated random number: Group I treated with valsartan (160 mg/d, n = 100), Group II amlodipine (10 mg/d, n = 100). Another 30 healthy subjects are enrolled as control group (Group III). Subjects in group I and II were asked to maintain their usual dietary and physical activity habits throughout the study. Treatment tolerability was assessed at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients, of both sexes with mild to moderate essential hypertension (diastolic blood pressure [DBP] >80 and ≤100 mmHg after a 2-week wash-out period, SBP systolic blood pressure>120 and 160 mmHg). Another 30 healthy subjects are enrolled as control group.

Exclusion Criteria:

* Subjects with age < 18 years and >65 years and those with two and more antihypertensive medications, those with diabetes, liver or kidney diseases, angina, myocardial infarction or stroke within 6 months, congestive heart failure, neurologic or psychiatric illness, secondary hypertension, known hypersensitivity to the drugs used in the study. also those with conditions that may have caused metabolic alterations within the past year (pregnancy, abdominal surgery, weight gain or loss of more than 3 kg) are excluded.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
LV mass index (g/m2) | three months
  Left ventricular mass index (LVMI) is a parameter used in echocardiography cardiac MRI.
  LVMI is calculated using the following equations:
  LVMI = LVM (left ventricular mass/body surface area left ventricular mass = 0.8{1.04[([LVEDD + IVSd +PWd]3 - LVEDD3)]} + 0.6 Where
  LVEDD = LV end-diastolic dimension (mm) IVSd = interventricular septal thickness at end-diastole (mm) PWd = posterior wall thickness at end-diastole (mm)
Concentration of Adiponectin (pg/ml) | three months
  Adiponectin is an adipocyte-secreted protein that circulates in the serum
Concentration of Leptin (ng/ml) | three months
  Leptin is a hormone secreted from fat cells that helps to regulate body weight.
Concentration of TNF-α (pg/ml) | Three months
  Tumor necrosis factor (TNF or TNF-α) is a major pro-inflammatory cytokine involved in early inflammatory events.
Concentration of hs-CRP (mg/L) | Three Months
  High sensitivity C-reactive protein a biomarker of inflammation and cardiovascular disease risk.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Werida, Ass. Prof., Study Director — Damanhour University
Locations (1):
- Tanta University Hospital, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tadic M, Cuspidi C, Ivanovic B, Ilic I, Celic V, Kocijancic V. Influence of White-Coat Hypertension on Left Ventricular Deformation 2- and 3-Dimensional Speckle Tracking Study. Hypertension. 2016 Mar;67(3):592-6. doi: 10.1161/HYPERTENSIONAHA.115.06822. Epub 2016 Jan 4. PMID 26729750
- [Background] Yilmaz MI, Sonmez A, Caglar K, Celik T, Yenicesu M, Eyileten T, Acikel C, Oguz Y, Yavuz I, Vural A. Effect of antihypertensive agents on plasma adiponectin levels in hypertensive patients with metabolic syndrome. Nephrology (Carlton). 2007 Apr;12(2):147-53. doi: 10.1111/j.1440-1797.2007.00764.x. PMID 17371337